CLINICAL TRIAL: NCT06727578
Title: A Pilot Assessment of the Safety and Efficacy of Pleural Irrigation for Retained Pleural Infection Using a Novel Irrigation Device
Brief Title: Pleural Irrigation With a Novel Devise.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Adnan Majid, MD, Chief, Section of Interventional Pulmonology, Division of Thoracic Surgery and Interventional Pulmonology, Beth Israel Deaconess Medical Center, Professor of Medicine, Harvard Medical School,, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000822
Record Dates: First submitted 2024-11-01; First posted 2024-12-11 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Pleural Effusion Disorder
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: of intrapleural saline irrigation with CLR irrigator

INTERVENTIONS:
Device: of intrapleural saline irrigation with CLR irrigator — patients will have a CLRTM port and CLRTM irrigator (CLR Medical, Calverton, MD, USA) added to their chest tube and atrium circuit to facilitate pleural irrigation.

SUMMARY:
Single-arm pilot trial of the use of intrapleural saline irrigation to treat retained pleural infections for patients with contraindications to standard of care intrapleural enzymatic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Retained pleural effusion identified via bedside ultrasound within the first 24 hours after chest tube insertion
* Patient is contraindicated from receiving intrapleural enzymatic therapy within the first 24 hours after chest tube insertion

Exclusion Criteria:

* Non-infectious cause of pleural fluid analysis findings listed above identified (e.g. malignancy)
* Post-procedural empyema or complicated parapneumonic effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic improvement (reduction in the ammount of pleural effusion messured in centimeters) by bed side ultrasound day 1,2,3,4,5. | Daily for 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies HE, Davies RJ, Davies CW; BTS Pleural Disease Guideline Group. Management of pleural infection in adults: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii41-53. doi: 10.1136/thx.2010.137000. No abstract available. PMID 20696693
- [Background] Gupta I, Eid SM, Gillaspie EA, Broderick S, Shafiq M. Epidemiologic Trends in Pleural Infection. A Nationwide Analysis. Ann Am Thorac Soc. 2021 Mar;18(3):452-459. doi: 10.1513/AnnalsATS.202001-075OC. PMID 33001756
- [Background] Sogaard M, Nielsen RB, Norgaard M, Kornum JB, Schonheyder HC, Thomsen RW. Incidence, length of stay, and prognosis of hospitalized patients with pleural empyema: a 15-year Danish nationwide cohort study. Chest. 2014 Jan;145(1):189-192. doi: 10.1378/chest.13-1912. No abstract available. PMID 24394842
- [Background] Grijalva CG, Zhu Y, Nuorti JP, Griffin MR. Emergence of parapneumonic empyema in the USA. Thorax. 2011 Aug;66(8):663-8. doi: 10.1136/thx.2010.156406. Epub 2011 May 26. PMID 21617169
- [Background] Light RW, Girard WM, Jenkinson SG, George RB. Parapneumonic effusions. Am J Med. 1980 Oct;69(4):507-12. doi: 10.1016/0002-9343(80)90460-x. PMID 7424940